CLINICAL TRIAL: NCT05161598
Title: PRE-APPROVAL ACCESS (PAA) Single Patient Request (SPR) TREATMENT GUIDELINES for Teclistamab (JNJ-64007957) for Treating Physician Use
Brief Title: Pre-approval Access Single Patient Request for Teclistamab (JNJ-64007957)
Status: No longer available | Type: Expanded Access
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108846; 64007957PTL4001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2021-12-03; First posted 2021-12-17 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Teclistamab — Teclistamab will be administered subcutaneously (SC).
  Other Names: JNJ-64007957

SUMMARY:
Teclistamab pre-approval access in relapsed or refractory multiple myeloma.

ELIGIBILITY:
Must have relapsed/refractory multiple myeloma (RRMM) and have evidence of disease progression after last therapy. Must have exhausted all available treatment options accessible as local standard of care (example. proteasome inhibitors [PIs], immunomodulatory imide drugs [IMIDs], anti CD38 monoclonal antibodies [mAbs] and therapies targeting Exportin 1 [XPO1] and B cell maturation antigen [BCMA]). Must not be eligible for a clinical trial with teclistamab or other medicines in this setting

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC